CLINICAL TRIAL: NCT03235284
Title: Efficacy of Nintendo WII and Exercises at Rehabilitation of Individuals With Parkinson's Disease: Randomized Clinical Trial
Brief Title: Nintendo WII and Exercises at Rehabilitation of Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, PIETRO ARAÚJO DOS SANTOS, Principal Investigator, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NintendoWii x Exercises
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease ande Video Games
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercises (Active Comparator): A program of therapeutic exercises (GC) based on the PNF method for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes. The GC treatment program consists of the following protocols: a) protocol 1: 20 minutes diagonal exercise upper limb (flexion-abduction-external rotation and extension-abduction-internal rotation),10 minutes diagonal exercise scapula (anterior and posterior elevation) and 10 minutes of exercise for trunk extension; b) protocol 2: 20 minutes diagonal exercise lower limb (flexion-abduction-external rotation and flexion-abduction-internal rotation),10 minutes diagonal exercise pelvis (anterior and posterior depression), and 10 minutes gait cycle training;
  Interventions: Other: Exercises
- Nintendo Wii (Active Comparator): Nintendo Wii program (GW) based on the use of the NW for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes.
  The GW treatment program consists of the following protocols: a) protocol 1 games (Boxing and Soccer); b) protocol 2 games (Golf and running). 20 minutes for each game
  Interventions: Other: Nintendo Wii
- Exercises and Nintendo Wii (Experimental): In GCW program will be performed 20 minutes GC protocol (1 or 2, used alternately between sessions a week) and 20 minutes GW protocol (1 or 2, used alternately between sessions a week), taking the time of the performed activities halved in both protocols
  Interventions: Other: Exercises and Nintendo Wii

INTERVENTIONS:
Other: Exercises — A program of therapeutic exercises (GC) based on the PNF method for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes. The GC treatment program consists of the following protocols: a) protocol 1: 20 minutes diagonal exercise upper limb (flexion-abduction-external rotation and extension-abduction-internal rotation),10 minutes diagonal exercise scapula (anterior and posterior elevation) and 10 minutes of exercise for trunk extension; b) protocol 2: 20 minutes diagonal exercise lower limb (flexion-abduction-external rotation and flexion-abduction-internal rotation),10 minutes diagonal exercise pelvis (anterior and posterior depression), and 10 minutes gait cycle training
  Arms: Exercises
Other: Nintendo Wii — Nintendo Wii program (GW) based on the use of the NW for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes.
  The GW treatment program consists of the following protocols: a) protocol 1 games (Boxing and Soccer); b) protocol 2 games (Golf and running). 20 minutes for each game
  Arms: Nintendo Wii
Other: Exercises and Nintendo Wii — In GCW program will be performed 20 minutes GC protocol (1 or 2, used alternately between sessions a week) and 20 minutes GW protocol (1 or 2, used alternately between sessions a week), taking the time of the performed activities halved in both protocols
  Arms: Exercises and Nintendo Wii

SUMMARY:
Patients with Parkinson's disease present motor dysfunctions such as stiffness, tremor, postural instability and bradykinesia, which leads to alterations of balance, necessitating specialized physiotherapeutic treatment. In this way this study aims to determine the effectiveness of two tools used in physiotherapy, kinesiotherapy and the Nintendo Wii. 45 patients will be evaluated through the Berg Balance Scale, Dynamic Gait Index, Timed up and go and PDQ-39, and will then be randomized to receive 16 sessions of Exercises or Nintendo Wii alone or together. After this period the patients will be reassessed to verify the effects of the techniques.

DETAILED DESCRIPTION:
Patients with Parkinson's disease present motor dysfunctions such as stiffness, tremor, postural instability and bradykinesia, which leads to alterations of balance, necessitating specialized physiotherapeutic treatment. In this way this study aims to determine the effectiveness of two tools used in physiotherapy, kinesiotherapy and the Nintendo Wii. 45 patients will be evaluated through the Berg Equilibrium Scale, Evaluated by the Dynamic Gait Index and the Timed up and go and PDQ-39. Later patients will be randomized to receive 16 sessions of Kinesiotherapy or Nintendo Wii alone or together, twice a week, for 50 minutes at the Neurociencias Outpatient Clinic of Teacher Magalhães Neto - FUBA. After this period the patients will be reassessed to verify the effects of the techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years,
* Stage 1 to 3 on the Hoehn and Yahr scale,
* Absence of visual or auditory impairment,

Exclusion Criteria:

* Presence of cognitive alterations according to MEEM: illiterate 19 points; 1 to 3 years of schooling 23 points; 4 to 7 years 24 points and above 7 years of 28 points
* Presence of other neurodegenerative diseases,
* Uncontrolled osteomioarticular or chronic diseases
* Participation in other rehabilitation programs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Complex Hospital Professor Edgard Santos, Federal University of Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: Related Info — http://dx.doi.org/10.4236/apd.2013.24018

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercises: The GC treatment program consists of the following protocols: a) protocol 1: 20 minutes diagonal exercise upper limb,10 minutes diagonal exercise scapula and 10 minutes of exercise for trunk extension; b) protocol 2: 20 minutes diagonal exercise lower limb ,10 minutes diagonal exercise pelvis, and 10 minutes gait cycle training;
- Nintendo Wii: Nintendo Wii program (GNW) based on the use of the NW for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes.
  The GNW treatment program consists of the following protocols: a) protocol 1 games (Boxing and Soccer); b) protocol 2 games (Golf and running). 20 minutes for each game
- Exercises and Nintendo Wii: Exercises and Nintendo Wii: A program of therapeutic exercises (GC) for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions). The GC treatment program consists of the following protocols: a) protocol 1 : 30 minutes diagonal exercise upper limb, 10 minutes diagonal exercise scapula and 20 minutes 20 minutes of extension exercises for the trunk; b) protocol 2: 20 minutes diagonal exercise lower limb,10 minutes diagonal exercise pelvis, and 10 minutes gait cycle training. Nintendo Wii program (GW) for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions). Protocol 1 games (Boxing e Soccer); b) protocol 2 games (Golf and Running). In GCW program will be performed 20 minutes G0 protocol (1 or 2, used alternately between sessions a week) and 20 minutes G1 protocol (1 or 2, used alternately between sessions a week), taking the time of the performed activities halved in both protocols.
Period: Overall Study
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii
Started | 15 | 15 | 15
Completed | 14 | 13 | 14
Not Completed | 1 | 2 | 1
Not completed — Adverse Event | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: patients with Parkinson's disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii | Total
Number analyzed (Participants) | 14 | 13 | 14 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 11
  >=65 years | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.8) | 61.7 (7.3) | 66.6 (8.2) | 64.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 10
  Male | 11 | 11 | 9 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 10 | 10 | 30
  White | 4 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Berg Balance Scale
Description: It is a scale that allows a functional assessment of the balance of the performance. It is based on 14 common items of everyday life, graduated from 0 to 4 points, reaching 56 points maximum score.
  It presents test reliability and re-test of 98%, another particularity of the scale is the non-linear relationship between the score and the risk of corresponding falls. The scores range from 0 to 56, the higher the score, the better the assessed individual's balance. Each point less on the scale corresponds to an increased risk of falls; between scores 56 to 54, each minus point is associated with a 3 to 4% increase in the risk of falls; between 54 and 46 an increase of 6 to 8% of chances for each point, being that below 36 points the risk of falls is almost 100%
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii
Number analyzed (Participants) | 14 | 13 | 14
Score on a scale
  Before | 40.5 (5.6) | 43.9 (5.3) | 41.6 (5.9)
  After | 45.6 (5.4) | 49.2 (4.4) | 47.1 (5.4)

2. Secondary Outcome: Dynamic Gait Index - DGI
Description: It is a scale that allows a functional assessment of the balance of the performance. Comprising 8 tasks with a score ranging from 0 to 3 points, maximum score of 24 points and minimum score of 0 points It consists of eight tasks involving walking in different sensory contexts, which include flat surface, change in gait speed, horizontal and vertical head movements, overpassing and bypassing obstacles, turning over the body axis itself, going up and down stairs . The maximum score is 24 points, and a score of 19 points or less predicts risk of falls. The scale has no gaps, only cutoff points. The higher the value, the better the gait performance. For patients with Parkinson's disease, values below 19 points predict major gait problems and high risk of falls.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii
Number analyzed (Participants) | 14 | 13 | 14
Units on a scale
  Before | 15.6 (4.7) | 15.7 (2.9) | 15.8 (1.9)
  After | 17.6 (3.6) | 19 (3.1) | 19.5 (2.2)

3. Secondary Outcome: Timed Up and Go - TUG
Description: The TUG measures, in seconds, the time it takes an individual to lift from a standard armchair (height of approximately 46 cm), walk a distance of 3 meters, turn, walk back to the chair and sit again.
  The patient is asked to lift from a chair (seat height of 45 cm and arms from 65 cm) to walk 3 meters, return and sit again, while the time spent in performing this task is timed.
  TUG up to ten seconds - individual without change of balance and with low risk of falls; (2) TUG between 11 and 20 seconds - individual with no significant alteration of balance, but presenting some fragility and medium risk of falls; (3) TUG greater than 20 seconds and less than 30 seconds - individual in need of intervention; (4) TUG greater than 30 seconds - individual at high risk for falls and with impaired mobility
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii
Number analyzed (Participants) | 14 | 13 | 14
Seconds
  Before | 10.7 (3.6) | 11.5 (5.1) | 13.9 (2.5)
  After | 8.2 (2.5) | 8.5 (2.1) | 10.6 (2.5)

4. Secondary Outcome: Parkinson's Disease Questionnaire (PDQ-39)
Description: 39 items divided into 8 domains. The total score ranges from 0 to 100, in which a lower score denotes a better perception of the patient's.
  It is divided into eight categories: mobility (10 items), daily life activities (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (3 items) and body discomfort (3 items) .43 The score ranges from 0 (no problem) to 100 (maximum problem level), ie low score indicates the individual's perception of a better quality of life .. These items can be grouped into three domains: physical, mental and social. The score is made by rule of three and transformed into values from 0 to 100, and higher values refer to poorer quality of life.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii
Number analyzed (Participants) | 14 | 13 | 14
Score on a scale
  Before | 32.7 [26.7 to 54] | 37.1 [24.5 to 45.3] | 32.9 [22.4 to 36.2]
  After | 25.7 [12.6 to 36.2] | 29.7 [22.4 to 35.1] | 23.5 [17.9 to 32.3]

ADVERSE EVENTS:
Time Frame: Two years
Groups:
- Exercises: A program of therapeutic exercises (GC) based on the PNF method for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes. The GC treatment program consists of the following protocols: a) protocol 1: 20 minutes diagonal exercise upper limb (flexion-abduction-external rotation and extension-abduction-internal rotation),10 minutes diagonal exercise scapula (anterior and posterior elevation) and 10 minutes of exercise for trunk extension; b) protocol 2: 20 minutes diagonal exercise lower limb (flexion-abduction-external rotation and flexion-abduction-internal rotation),10 minutes diagonal exercise pelvis (anterior and posterior depression), and 10 minutes gait cycle training. Fatigue, fainting, or changes in blood pressure may occur.
- Nintendo Wii: Nintendo Wii program (GW) based on the use of the NW for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes.
  The GW treatment program consists of the following protocols: a) protocol 1 games (Boxing and Soccer); b) protocol 2 games (Golf and running). 20 minutes for each game. Fatigue, fainting, or changes in blood pressure may occur.
- Exercises and Nintendo Wii: A program of therapeutic exercises (GC) for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions). The GC treatment program consists of the following protocols: a) protocol 1 : 30 minutes diagonal exercise upper limb, 10 minutes diagonal exercise scapula and 20 minutes 20 minutes of extension exercises for the trunk; b) protocol 2: 20 minutes diagonal exercise lower limb,10 minutes diagonal exercise pelvis, and 10 minutes gait cycle training. Nintendo Wii program (GW) for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions). Protocol 1 games (Boxing e Soccer); b) protocol 2 games (Golf and Running). In GCW program will be performed 20 minutes G0 protocol (1 or 2, used alternately between sessions a week) and 20 minutes G1 protocol (1 or 2, used alternately between sessions a week), taking the time of the performed activities halved in both protocols. Fatigue, fainting, or changes in blood pressure
Arm/Group | Exercises | Nintendo Wii | Exercises and Nintendo Wii
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
The absence of an instrument to verify the presence of depression, which is a clinical condition present in some patients with PD and may have influenced the absence of more significant results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03235284/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03235284/ICF_001.pdf